CLINICAL TRIAL: NCT04926623
Title: Multicenter, Open-label, Randomized Trial to Compare the Effectiveness of Structured Education and Safety of FreeStyle Libre or Self-Monitoring of Blood Glucose (SMBG) in Patients With Type 2 Diabetes Mellitus Using Multiple Daily Injections or Insulin Pumps
Brief Title: Freestyle Libre-based Education on MDI in T2DM (FreEdoM-2)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DWFSL-P401
Record Dates: First submitted 2021-06-10; First posted 2021-06-15 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CGM with Structured Education (Experimental): CGM with Structured Education
  Interventions: Device: FreeStyle Libre 24 weeks
- CGM with Standard Education (Active Comparator): CGM with Standard Education
  Interventions: Device: FreeStyle Libre 24 weeks
- SMBG with Standard Education (Active Comparator): SMBG and CGM with Standard Education
  Interventions: Other: SMBG (22 weeks) and blind CGM (2 weeks)

INTERVENTIONS:
Device: FreeStyle Libre 24 weeks — FreeStyle Libre flash sensor-based glucose monitoring system (FSGM; Abbott Diabetes Care, Witney, Oxon, UK)
  Arms: CGM with Standard Education; CGM with Structured Education
Other: SMBG (22 weeks) and blind CGM (2 weeks) — Self-Monitoring of Blood Glucose and Continuous Glucose Monitoring
  Arms: SMBG with Standard Education

SUMMARY:
Multicenter, Open-label, Randomized Trial to Compare the Effectiveness of Structured Education and Safety of FreeStyle Libre or Self-Monitoring of Blood Glucose (SMBG) in patients with type 2 Diabetes Mellitus using Multiple Daily Injections or Insulin Pumps

DETAILED DESCRIPTION:
All subjects must participate in Blind Continuous Glucose Monitoring(CGM) for two weeks prior to Visit 2 visit (random assignment).

Subjects who meet the selection/exclusion criteria in Visit 2 visits are randomly assigned to the test group (personal in-depth education and FreeStyle Libre) or control 1 (standard education and FreeStyle Libre) or control 2 (standard education and SMBG) at a 1:1:1 ratio.

In the test group, personal in-depth education is conducted at baseline (Visit 2), 4 weeks (Visit 3), 8 weeks (Visit 4), 12 weeks (Visit 5), and 18 weeks (Visit 6), and the time required for education and preparation time required for patient education are checked.

Control groups 1 and 2 conduct routine insulin basic injection training as standard education at baseline (Visit 2) and 12 weeks (Visit 5).

After randomization, FreeStyle Libre is applied to the test group and control group 1 for 24 weeks, and SMBG is performed for 22 weeks and Blind CGM is applied for 2 weeks at 22 weeks (Visit 7).

Blood glucose measurements collected from FreeStyle Libre are collected through the reader program, and are checked in real time by researchers and used for education, research, and analysis. Prior to the implementation of FreeStyle Libre for the collection of real-time blood sugar collected through FreeStyle Libre, the subject is given consent to disclose blood sugar information.

All subjects visit baseline (Visit 2), 12 weeks (Visit 5), and 24 weeks (Visit 8) to conduct surveys on physical examinations, blood tests and urine tests (Central Lab), and treatment satisfaction questionnaire (DTSQ).

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes patients aged 19 and under 75 years.
2. Multiple insulin injections at the time of screening (at least one base insulin and two or more fast-acting insulin. However, one insulin aspart/insulin degludec + one insulin aspart or two or more insulin aspart/insulin degludec can be included.) or those who have been using an insulin pump for at least 12 weeks.
3. HbA1c of not less than 7.5% and not more than 12.0% at the time of screening
4. patients who agree to use FreeStyle Libre for medical care and research
5. patients who voluntarily signed a written consent form

Exclusion Criteria:

1. Those who have difficulty in education due to severe systemic diseases (e.g., terminal renal failure requiring dialysis, cirrhosis above Child-Pugh Class C), cognitive impairment, and mental illness.
2. Those who are taking drugs that may affect metabolism per screening time (e.g., adrenocortical hormones, immunosuppressants, etc.) (However, those who have taken the same dose for more than 12 weeks until screening time and who are not scheduled to change drug dose can participate in this study.)
3. Those with clinically significant cardiovascular diseases (heart failure, angina, myocardial infarction, cerebral infarction, etc.) within 24 weeks of screening.
4. Those who have a glomerular filtration rate (eGFR) of <15 mL/min.
5. A person with severe diabetes complications that deteriorate or newly occur within 3 months of screening and require emergency treatment.
6. Pregnant or lactating persons.
7. Pregnancy is planned during the study period, effective contraception (if condoms, oral contraceptives, intrauterine contraceptives, injections, transplants, contraceptives, or absolute abstinence, such as periodic abstinence (e.g., Krenda, ovulation, symptom body temperature) and resection are not considered as recognized contraceptives) for women or men.
8. Those who find other researchers inappropriate for participation in research.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2021-06-17 (Actual); Primary Completion 2022-10-26 (Actual); Study Completion 2023-04-04 (Actual)

PRIMARY OUTCOMES:
HbA1c (%) changes | 24 weeks
  HbA1c (%) changes at 24 weeks compared to baseline

SECONDARY OUTCOMES:
HbA1c (%) changes | 12 weeks
  HbA1c (%) changes at 12 weeks compared to baseline
Percentage of time in level 2 hypoglycemia (<54 mg/dL) | 24 weeks
  Percentage of time in level 2 hypoglycemia (<54 mg/dL) at 24 weeks compared to baseline
Percentage of time in level 1 hypoglycemia (<70- 54 mg/dL) | 24 weeks
  Percentage of time in level 1 hypoglycemia (<70- 54 mg/dL) at 24 weeks compared to baseline
Percentage of time in level 1 hypoglycemia (> 180 mg/dL) | 24 weeks
  Percentage of time in level 1 hypoglycemia (> 180 mg/dL) at 24 weeks compared to baseline
Percentage of time in level 2 hypoglycemia (> 250 mg/dL) | 24 weeks
  Percentage of time in level 2 hypoglycemia (> 250 mg/dL) at 24 weeks compared to baseline
Percentage of time in range (70 - 180mg/dL) | 24 weeks
  Percentage of time in range (70 - 180mg/dL) at 24 weeks compared to baseline
Mean glucose changes | 24 weeks
  Mean glucose changes at 24 weeks compared to baseline
Coefficient of variation(CV) changes | 24 weeks
  Coefficient of variation(CV) changes at 24 weeks compared to baseline
Diabetes Treatment Satisfaction Questionnaire (DTSQ) changes | 12 weeks
  Diabetes Treatment Satisfaction Questionnaire (DTSQ) changes at 12 weeks compared to baseline
Diabetes Treatment Satisfaction Questionnaire (DTSQ) changes | 24 weeks
  Diabetes Treatment Satisfaction Questionnaire (DTSQ) changes at 24 weeks compared to baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kim JY, Jin SM, Sim KH, Kim BY, Cho JH, Moon JS, Lim S, Kang ES, Park CY, Kim SG, Kim JH. Continuous glucose monitoring with structured education in adults with type 2 diabetes managed by multiple daily insulin injections: a multicentre randomised controlled trial. Diabetologia. 2024 Jul;67(7):1223-1234. doi: 10.1007/s00125-024-06152-1. Epub 2024 Apr 19. PMID 38639876